CLINICAL TRIAL: NCT00002278
Title: 28 Day Protocol for the Treatment of Cryptosporidiosis in AIDS Patients With Diclazuril (R64,433)
Brief Title: A 28-Day Study of Diclazuril in the Treatment of Cryptosporidiosis in Patients With AIDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Janssen, LP (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 038B; JRD 64,433/1102
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1990-07

CONDITIONS: Cryptosporidiosis; HIV Infections
Keywords: AIDS-Related Opportunistic Infections; Cryptosporidiosis; Diarrhea; diclazuril; Coccidiostats; Acquired Immunodeficiency Syndrome
MeSH Terms: conditions — Cryptosporidiosis; HIV Infections; AIDS-Related Opportunistic Infections; Diarrhea; Acquired Immunodeficiency Syndrome | interventions — diclazuril

INTERVENTIONS:
Drug: Diclazuril

SUMMARY:
To evaluate the safety and efficacy of diclazuril capsules as a treatment for cryptosporidial related diarrhea in AIDS patients who have been treated in the double-blind study # JRD 64,433/1101 and have relapsed, or de-novo patients who have been diagnosed with cryptosporidial related diarrhea and who meet the inclusion and exclusion criteria of this protocol.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Zidovudine (AZT).
* Didanosine (ddI) allowed but discouraged, must have been stabilized on a constant dose for 3 weeks or more.
* Aerosolized pentamidine.
* Nystatin for control of oropharyngeal infections. Nystatin must not be taken within two hours of diclazuril.
* Ganciclovir therapy only for CMV retinitis is permitted if the patient has been treated for at least 4 weeks prior to study entry and is stable on the drug.
* Loperamide may be taken if patient has been on long term loperamide prior to study entry but should not be started during the course of this protocol.

Patients must have the following:

Written informed consent given after the purpose and nature of the study, as well as the possible adverse effects related to the study drug, have been explained.

* Be willing and able to return for all subsequent weekly visits and the two week visit post completion of therapy (follow-up).

Prior Medication:

Allowed:

* Diclazuril.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Uncontrolled vomiting.
* Estimated survival less than 28 days.
* Other treatable enteric pathogens must be treated and eradicated prior to study entry.

Concurrent Medication:

Excluded:

* Amphotericin B.
* Other antibiotics or antiprotozoal drugs.
* Other investigational agents.
* Trimethoprim/sulfamethoxazole.
* Antifungal medications except nystatin.
* Ganciclovir for other than Cytomegalovirus (CMV) retinitis.
* Antidiarrheal agents other than patients on long term loperamide prior to study entry.

Patients with the following are excluded:

* Undependable in following the instructions of the investigator.
* Not able to swallow capsules.
* Uncontrolled vomiting.
* Estimated survival less than 28 days.

Prior Medication:

Excluded:

* Diclazuril within 2 weeks of study entry.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Cornell Univ Med Ctr, New York, New York
  - Saint Luke's - Roosevelt Hosp Ctr, New York, New York